CLINICAL TRIAL: NCT05258656
Title: Childhood Activities Nutrition and Development Oversight
Acronym: CANDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Food Allergy Research & Education (Other)
Responsible Party: Principal Investigator, Ruchi Gupta, Professor of Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-4156
Record Dates: First submitted 2022-02-11; First posted 2022-02-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Environmental Exposure
Keywords: infant development; health promotion
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive education about nutrition, resources, and specific instructions on promoting healthy development of their infant, including guidance regarding infant sleep, screen time, and building healthy relationships.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): The control group will receive specific instructions on promoting healthy development of their infant, including guidance regarding infant sleep, screen time, and building healthy relationships.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive education about nutrition, resources, and specific instructions on promoting healthy development of their infant, including guidance regarding infant sleep, screen time, and building healthy relationships.
  Arms: Intervention
Behavioral: Control — The control group will receive specific instructions on promoting healthy development of their infant, including guidance regarding infant sleep, screen time, and building healthy relationships.
  Arms: Control

SUMMARY:
The overall goal of this study is to understand how common conditions in childhood develop and if by providing specific health education and resources to parents/caregivers we can promote healthy development. This study will provide information and instruction on several aspects of infant care including, sleep, nutrition, building a healthy relationship with your baby, and healthy screen time use.

DETAILED DESCRIPTION:
This study is a randomized controlled trial that will recruit parents/caregivers and infants infants living in the Greater Chicago area . The study will follow these infants until they are three years old.

The intervention arm will receive education about nutrition, resources, and specific instructions on feeding and caring for their infants. The control arm will receive education about infant development and helpful tips about infant sleep, screen time, and building healthy relationships. In addition, all caregivers will be asked to fill out surveys and come to research visits during the study period. There will be a total of 4 study visits during the three years of the study. There will be optional blood, stool, and skin testing of the child at each study visit. Two visits will take place during the first year of life, followed by visits around the child's 2nd and 3rd birthdays.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian(s) must understand and provide informed consent
* Infant <26 weeks of age at enrollment
* Willing to be randomized to either intervention or control
* In good general health as evidenced by medical history
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Child assigned male or female sex at birth

Exclusion Criteria:

* Infant completed less than 28 weeks gestation
* Co-morbid medical diagnoses that would prevent caregivers from initiating solid foods per protocol, such as dysphagia, chronic aspiration, malformations, etc.
* Co-morbid medical diagnoses that would require specialized diet/nutritional needs, such as congenital heart disease, genetic/metabolic disorders, malignancy, etc.
* Caregivers who express unwillingness to introduce peanut, milk, egg, or cashew
* Caregivers who cannot provide informed consent in English or Spanish
* Parents planning to move away from study sites before child is 12 months of age
* Investigator or designee considers that the participant or parent/guardian would be unsuitable for inclusion in the study
* Infant with a sibling enrolled in the study

Max Age: 26 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
One year Assessment | ≈12 months of age
  Caregivers and their child will be asked to attend a research study visit with a physician around the child's 1st birthday that may involve brief examination of the child's skin, surveys about the child's medical history and diet, a supervised feeding of certain common foods, and/or collection of a blood sample.

SECONDARY OUTCOMES:
Two year assessment | ≈24 months of age
  Caregivers and their child will be asked to attend a research study visit with a physician around the child's 2nd birthday that may involve brief examination of the child's skin, surveys about the child's medical history and diet, a supervised feeding of certain common foods, and/or collection of a blood sample.
Three year assessment | ≈36 months of age
  Caregivers and their child will be asked to attend a research study visit with a physician around the child's 3rd birthday that may involve brief examination of the child's skin, surveys about the child's medical history and diet, a supervised feeding of certain common foods, and/or collection of a blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchi S Gupta, MD MPH, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
We plan to share deidentified, limited data sets and corresponding analytic code with other researchers following the publication of the study data. The protocol, Statistical Analysis Plan, and Informed Consent Forms will also be published online as supplemental appendices and will be made available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and supporting information will be available indefinitely upon their publication.
Access Criteria: Published study datasets will be publicly available.
  Requests for unpublished data will be reviewed by the PI and advisory board and approved if deemed to have scientific merit.